CLINICAL TRIAL: NCT05003518
Title: ParentText User Engagement and Effectiveness Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient participants were recruited for the optimisation trial. Study procedures revised to conduct a pilot of intervention acceptability, feasibility, and preliminary change in psychosocial behavioural outcomes.
Sponsor: University of Oxford (Other)
Collaborators: IDEMS International (Unknown); UNICEF South Africa (Unknown); UNICEF Malaysia (Unknown); UNICEF Sri Lanka (Unknown); UNICEF Jamaica (Unknown); UNICEF Philippines (Unknown); Health Promotion Bureau, Sri Lanka (Unknown); Universiti Putra Malaysia (Other); Ateneo de Manila University (Other); University of Cape Town (Other); The LEGO Foundation (Unknown)
Responsible Party: Principal Investigator, DrJamieLachman, Senior Research and Teaching Fellow, University of Oxford
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: ParentTextOpti
Record Dates: First submitted 2021-07-28; First posted 2021-08-12 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Engagement; Positive Parenting; Child Maltreatment; Intimate Partner Violence
Keywords: Engagement; Chatbot; Digital Behaviour Change Intervention; Parenting Intervention; Optimisation; Positive Parenting; Child Maltreatment; Intimate Partner Violence

STUDY DESIGN:
Intervention Model Description: A factorial design will be used testing the four components, with a total of 16 conditions. The purpose of this factorial experiment is to estimate the main effects of the four intervention components and interactions between the components, not to compare the 16 experimental conditions to each other.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- Condition 1: Low Personalisation+Low Frequency (Experimental): The intervention will have low levels of personalisation and one message a day will be sent to participants.
  Interventions: Behavioral: ParentText
- Condition 2: High Personalisation+Low Frequency (Experimental): The intervention will have high levels of personalisation (utilise the user's nickname and their child's nickname) and one message a day will be sent to participants.
  Interventions: Behavioral: ParentText
- Condition 3: Low Personalisation+High Frequency (Experimental): The intervention will have low levels of personalisation and three messages a day will be sent to participants.
  Interventions: Behavioral: ParentText
- Condition 4: High Personalisation+High Frequency (Experimental): The intervention will have high levels of personalisation and three messages a day will be sent to participants.
  Interventions: Behavioral: ParentText
- Condition 5: High Personalisation+Low Frequency+Gamification (Experimental): The intervention will have high levels of personalisation (utilise the user's nickname and their child's nickname), contains gamified progress updates, and one message a day will be sent to participants.
  Interventions: Behavioral: ParentText
- Condition 6: Low Personalisation+High Frequency+Gamification (Experimental): The intervention will have low levels of personalisation, contains gamified progress updates, and three messages a day will be sent to participants.
  Interventions: Behavioral: ParentText
- Condition 7: High Personalisation+High Frequency+Gamification (Experimental): The intervention will have high levels of personalisation (utilise the user's nickname and their child's nickname), contains gamified progress updates, and three message a day will be sent to participants.
  Interventions: Behavioral: ParentText
- Condition 8: Low Personalisation+Low Frequency+Gender Targeting (Experimental): The intervention will have low levels of personalisation, contains gender targeted messages, and one message a day will be sent to participants.
  Interventions: Behavioral: ParentText
- Condition 9: High Personalisation+Low Frequency+Gender Targeting (Experimental): The intervention will have high levels of personalisation (utilise the user's nickname and their child's nickname), contains gender targeted messages, and one message a day will be sent to participants.
  Interventions: Behavioral: ParentText
- Condition 10: Low Personalisation + High Frequency + Gender Targeting (Experimental): The intervention will have low levels of personalisation, contains gender targeted messages, and three message a day will be sent to participants.
  Interventions: Behavioral: ParentText
- Condition 11: High Personalisation + High Frequency + Gender Targeting (Experimental): The intervention will have high levels of personalisation (utilise the user's nickname and their child's nickname), contains gender targeted messages, and three message a day will be sent to participants.
  Interventions: Behavioral: ParentText
- Condition 12: Low Personalisation + Low Frequency + Gamification + Gender Targeting (Experimental): The intervention will have low levels of personalisation, contains gender targeted messages and gamified progress updates. Participants will be sent one message a day.
  Interventions: Behavioral: ParentText
- Condition 13: High Personalisation + Low Frequency + Gamification + Gender Targeting (Experimental): The intervention will have high levels of personalisation (utilise the user's nickname and their child's nickname), contains gender targeted messages and gamified progress updates. Participants will be sent one message a day.
  Interventions: Behavioral: ParentText
- Condition 14: Low Personalisation + High Frequency + Gamification + Gender Targeting (Experimental): The intervention will have low levels of personalisation (utilise the user's nickname and their child's nickname), contains gender targeted messages and gamified progress updates. Participants will be sent three message a day.
  Interventions: Behavioral: ParentText
- Condition 15: High Personalisation + High Frequency + Gamification + Gender Targeting (Experimental): The intervention will have high levels of personalisation (utilise the user's nickname and their child's nickname), contains gender targeted messages and gamified progress updates. Participants will be sent three messages a day.
  Interventions: Behavioral: ParentText
- Condition 16: Low Personalisation+Low Frequency+Gamification (Experimental): The intervention will have low levels of personalisation (utilise the user's nickname and their child's nickname), contains gamified progress updates, and one message a day will be sent to participants.
  Interventions: Behavioral: ParentText

INTERVENTIONS:
Behavioral: ParentText — ParentText delivers content, aligning with children's developmental stages (0-23 months, 2-9 years, 10-17 years). ParentText content is delivered through text messages, images, audio and video for parents/ caregivers and their children. Parents receive parenting content surrounding three themes: 1) relationship building by spending time together, 2) positive reinforcement, 3) stress reduction for parents and caregivers. Further supportive content is available for parents of children living with disabilities, child development, online child safety, talking about COVID-19 with children, family budgeting, family harmony, helping with schoolwork and sexual violence prevention.

SUMMARY:
The study has two main aims. The first aim is to optimise user engagement in ParentText. The goal is to identify the optimal delivery of ParentText for parents/caregivers from low- and middle-income countries, using a randomised between-subjects factorial experimental design.

The second aim is to examine the preliminary effectiveness of the chatbot adaption of the Parenting for Lifelong Health programme, ParentText, on the primary outcome of child maltreatment and secondary outcomes of positive parenting, parental self-efficacy, parental communication about sexual abuse, financial stress, parental stress, child behaviour problems, and intimate partner violence.

This study is part of a multi-phase research project. The full research project has been registered to the Open Science Framework platform.

To address the first aim, the investigators will be conducting a factorial experiment which will examine the impact of four components, Personalisation (High/Low), Gamification (On/Off), Gender Targeting (On/Off), Frequency of message (1 per day/ 3 per day) on participant engagement. The factorial experiment will be conducted in two countries, Malaysia and South Africa. Within each country, the investigators have local partners who will be involved in deploying the intervention and recruiting participants. Parents/caregivers will be primarily recruited through country-specific UNICEF U-Report platforms and government partners. RapidPro, the programme on which the chatbot is deployed, will randomly allocate participants to the 16 experimental conditions. The purpose of the factorial experiment is to estimate the main and interaction effects of the four components. Based on the results the investigators will optimise the delivery of ParentText by selecting components or components levels that promote the highest level of engagement based on effect size.

The second aim will be addressed by conducting latent growth curve models or multi-level models, to examine the changes in outcome variables over time. The experiment will be conducted across five countries, Malaysia, South Africa, the Philippines, Jamaica and Sri Lanka. Within each country, the investigators have local partners who will be involved in deploying the intervention and recruiting participants.

DETAILED DESCRIPTION:
Research has shown that the modification of parenting programmes from being held in-person to being delivered digitally has been successful. Meta-analytic and systematic reviews carried out in HMICs have illustrated that digital parenting interventions have similar effect sizes to in-person interventions. Although these results are promising, there are few gaps within the literature that have not been addressed. First, the majority of research is being conducted in High-Income Countries (HICs). Therefore, results cannot be generalised to LMICs, where differences in context and culture could have an impact on the effectiveness of digital parenting interventions. Second, parenting interventions are deployed on a variety of different technological platforms, however, a limited amount of research has focused on examining emerging platforms, with the focus primarily being on app or internet-based interventions. Therefore little is known in regards to the effectiveness of more novel intervention platforms, such as chatbots.

Whilst the digitalisation of parenting programmes allows for the widespread dissemination and utilisation of the intervention, engagement rates for digital interventions remain low. Engagement with digital behaviour change interventions can be described as the extent (e.g. amount, frequency, duration, depth) of usage, and as a subjective experience characterised by attention, interest and affect. Low engagement compromises the effectiveness of parenting programmes, as the user is required to enrol and engage with the intervention for the programme to have an influence on behaviour. Intervention developers have begun employing technological platforms, such as chatbots, that are designed with the intention to overcome low user engagement rates.

Parenting research investigating digital intervention components which facilitate engagement remains scarce. Broadening the scope beyond the field of parenting, reviews of quantitative and qualitative research examining digital behaviour change interventions, identified an assortment of behaviour change techniques and persuasive system design principles which have been found to facilitate and impede engagement and effectiveness. However, few consistent patterns emerged regarding what techniques and principles consistently facilitate engagement and effectiveness, and for whom. There is a requirement for the isolated techniques and principles utilised within digital parenting interventions to be tested, to identify which intervention components influence engagement and intervention effectiveness and apply this research to optimise parenting interventions.

The first aim of this study is to optimise user engagement in ParentText and to identify the optimal delivery of ParentText for parents/caregivers from low- and middle-income countries. The investigators will be addressing three research questions:

1. How do different component levels impact ParentText user engagement and retention in terms of a) message personalisation (high/low), b) gendered targeted messages (on/off), c) gamification of module completions (on/off) and d) frequency of messages (high/low)?
2. Are there any interaction effects between different component levels of ParentText on user engagement and retention?
3. How does the effectiveness of each component or component level on user engagement vary by different population characteristics (i.e., parent/child age and gender, parent/caregiver marital status, parent/caregiver relationship to the child, and experience of COVID-19)?

The factorial experiment will be conducted across two countries, Malaysia and South Africa. Within each country, the investigators have local partners who will be involved in deploying the intervention and recruiting participants who take care of a child aged between 0 and 17 years old. Parents/caregivers will be primarily recruited through country-specific UNICEF U-Report platforms and government partners.

The following components have been selected, based on research that concluded that these components have been efficient in increasing engagement with digital interventions.

Component A: Personalisation (High/Low): Half of the participants will receive high levels of personalisation, receiving messages that utilise their (nick)name and the child's (nick)name. Half of the participants will not receive this type of personalisation.

Component B: Gendered Targeted Messages (On/Off): Half of the participants will receive messages that are tailored towards either being a female or male caregiver. The other half will not.

Component C: Gamification of Module Completion (On/Off): Half of the participants will receive a gamified progress update on what modules that they have completed. This will be represented as the House of Support. As the parent completes parenting skills, the layers of the house will fill in, representing their progress. The other half of the participants will not be receiving gamified progress updates.

Component D: Frequency of Messages (High/Low). Half of the participants will receive 3 interactions a day (high intensity), the other half will receive 1 interaction a day (low intensity).

The current factorial experimental trial will randomise participants into the 16 experimental conditions. Although this experiment has 16 experimental conditions, it is not a 16-arm RCT. The purpose of this factorial experiment is to estimate the main and intervention effects between the components and not to compare them to one another.

The study will examine the following hypotheses:

Hypotheses

* Participants who receive high levels of personalisation will show higher levels of engagement in ParentText, than compared to users receiving low levels of personalisation.
* Participants who receive gender-targeted messages will show higher levels of engagement in ParentText, than compared to users receiving no gender-targeted messages.
* Participants who receive gamified progress updates will show higher levels of engagement in ParentText, than compared to users receiving non-gamified progress updates.

Exploratory Hypotheses

* The investigators will explore how the frequency of messages will impact engagement.
* The investigators will explore how the effectiveness of components on engagement will vary dependent on demographic characteristics.
* The investigators will explore interaction effects between experimental components.

The second aim of the study is to examine the preliminary effectiveness of the chatbot adaption of the Parenting for Lifelong Health programme, ParentText on the primary outcome of child maltreatment and the secondary outcomes of positive parenting, parental self-efficacy, parental communication about sexual abuse, financial stress, parental stress, child behaviour problems, IPV, attitudes toward gender roles and IPV, and gender-equitable behaviours. The investigators will be investigating five research questions:

1. How does overall child maltreatment (primary outcome) change over time for parents/caregivers engaged in the ParentText intervention?
2. How do the following secondary outcomes change over time for parents/caregivers engaged in the ParentText intervention: physical abuse, emotional abuse, positive parenting, parental self-efficacy, parental communication about sexual abuse, financial stress, parental stress, child behaviour problems, intimate partner violence (IPV) victimisation and perpetration, attitudes toward intimate partner violence (IPV) and gender roles, and gender-equitable behaviours?
3. How do changes in secondary outcomes mediate change in overall child maltreatment?
4. How do changes in primary and secondary outcomes vary based on different population characteristics (i.e., parent/child age and gender, parent/caregiver marital status, parent/caregiver relationship to the child, and experience of COVID-19)?
5. What is the association between user engagement and change over time in primary outcomes and secondary outcomes?

Exploratory Hypotheses

* ParentText will have a significant impact on our primary outcome, decreasing child maltreatment.
* ParentText will have a significant impact on our secondary outcomes, increasing positive parenting, parental self-efficacy, parental communication about sexual abuse, gender-equitable behaviours and improving attitudes toward gender roles and IPV, as well as reducing financial stress, parental stress, child behaviour problems, intimate partner violence (IPV) victimisation and perpetration.
* The investigators will explore how the impact of ParentText will vary depending on user engagement and demographic characteristics.
* The investigators will also explore interaction effects between experimental components.

The experiment will be conducted in five countries, Malaysia, South Africa, Jamaica, the Philippines and Sri Lanka. Country specific recruitment is outlined below:

South Africa: Investigators will collaborate with Clowns Without Borders South Africa and the Department of Social Development to deploy and recruit participants in the Northern Cape. Participants will be recruited by radio announcements. The investigators are also collaborating with UNICEF South Africa who will assist in recruiting participants over the age of 20 via their U-Report Platform (N = 79,800). UNICEF South Africa will send U-reporters an unsolicited recruitment message that is accompanied by a link that takes users to the landing site of ParentText.

Malaysia: 20-35 participants will be recruited by our implementing partner, Generasi Gemilang from their family programmes. Participants will also be recruited either by UNICEF via their U-Report Platform (N = 25,200) or through the National Population and Family Development Board (LPPKN), which will blast messages to individuals who have previously participated in the LPPNK parenting workshops (N = 20,000).

Jamaica: Participants will be recruited in collaboration with UNICEF Jamaica and Parenting Partners Caribbean as part of the Spotlight Initiative, a community-wide intervention aimed at reducing violence against women and girls. Participants will be recruited in four parishes (N = 1,000). Parents and caregivers from the Spotlight initiative will be recruited by community youth activists, leaflets, radio announcements, posters, and other community-wide activities.

The Philippines: Participants will be recruited in collaboration with the Philippine Department of Social Welfare and Development. 30 families will be targeted who are enrolled in a conditional cash transfer programme (4Ps) who live in the Valenzuela municipality of Metro Manila.

Sri Lanka: Participants will be recruited in collaboration with the Health Promotion Bureau. Over 492,640 people follow this channel. The population includes media personal, health care service providers, community leaders, employers at all levels of industry and their organisations: hotels, supermarkets, banks, Ceylon Employer's Federation and the general public who uses Viber social media in Sri Lanka. The Health Promotion Bureau will select randomly individuals who are over 18 to receive a recruitment message to ParentText.

ELIGIBILITY:
Inclusion criteria for the participating parents/caregivers: over 18 years old, currently caring for a child between the ages of 0 to 17 years, access to a phone which can either receive SMS or has access to internet, and has provided consent to participate in the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1400 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Overall response to ParentText messages | Through study completion, an average of 16 weeks
  Number of many messages the participants responded to or timed out from the intervention (no engagement for 2 hours or more). This is a measure of engagement with the chatbot.
Overall completion rate of ParentText Content | Through study completion, an average of 16 weeks
  Number of the overall content the participant completed. This is a measure of completion of the programme.
Change over time in Child Maltreatment | Through study completion, an average of 16 weeks
  Child maltreatment will be a composite measure utilising two items adapted from the reduced version of the ISPCAN Child Abuse Screening Tool-Trial Parent Version (ICAST-TP) (Meinck et al., 2018), which is adapted from the survey instrument ICAST-Parent Version (ICAST-P) (Runyan et al., 2009). The ICAST-P was developed to be deployed multi-nationally and multi-culturally and has been successfully utilised in LMICs (Nøkleby et al., 2019). The ICAST-TP measures parental reports of incidences of abuse perpetrated against their child over the past week and asks parents/caregivers to answer a frequency score on a scale of 0 to 7 times. One item will assess physical abuse, "How many days in the past week did you physically discipline your children by hitting, spanking, or slapping with your hand or an object like a stick or a belt?". The other item will assess emotional abuse, "How many days in the past week did you shout, scream, or yell at your children?".

SECONDARY OUTCOMES:
Rate of response to tip offers | Through study completion, an average of 16 weeks
  This is a measure of engagement with the chatbot parenting content messages.
Rate of response to calm messages | Through study completion, an average of 16 weeks
  This is a measure of engagement with the chatbot stress-reduction messages.
Rate of response to praise messages | Through study completion, an average of 16 weeks
  This is a measure of engagement with the chatbot positive reinforcement messages.
Rate of response to supportive messages | Through study completion, an average of 16 weeks
  This is a measure of engagement with the chatbot supportive messages.
Rate of response to check in messages | Through study completion, an average of 16 weeks
  This is a measure of engagement with the chatbot check-in messages.
The number of messages the participant sent to the chatbot within a parenting skill. | Through study completion, an average of 16 weeks
  This is a measure of engagement with the programme.
The completion rate of parenting tips | Through study completion, an average of 16 weeks
  This is a measure of completion of the parenting modules during the programme.
The completion rate of self-led content | Through study completion, an average of 16 weeks
  This is a measure of completion of on-demand content during the programme.
The completion rate of survey assessments | Through study completion, an average of 16 weeks
  This is a measure of completion of assessment tools.
The completion rate of home practice | Through study completion, an average of 16 weeks
  This is a measure of engagement with applying parenting skills learned through the chatbot.
Experience with the skill | Through study completion, an average of 16 weeks
  This is a measure of the participants experience with engaging with the skill.
Consent to survey | Through study completion, an average of 16 weeks
  Participants can respond yes, no, or timeout to giving consent to the survey. This is a measure of engagement with the survey.
Response to survey questions | Through study completion, an average of 16 weeks
  Participants can respond, skip, or timeout to survey questions. This is a measure of engagement with the survey.
Participant Active Dropout | Through study completion, an average of 16 weeks
  Participants that actively exit the intervention.
Participant Passive Dropout | Through study completion, an average of 16 weeks
  Participants who timeout of the intervention and do not reengage with the intervention after one week.
Change over time in Physical Abuse | Through study completion, an average of 16 weeks
  Physical abuse will be assessed using one item adapted from the reduced version of the ISPCAN Child Abuse Screening Tool-Trial Parent Version (ICAST-TP) (Meinck et al., 2018). The item will assess physical abuse by asking, "How many days in the past week did you physically discipline your children by hitting, spanking, or slapping with your hand or an object like a stick or a belt?"
Change over time in Emotional Abuse | Through study completion, an average of 16 weeks
  Emotional abuse will be assessed using an item adapted from the reduced version of the ISPCAN Child Abuse Screening Tool-Trial Parent Version (ICAST-TP) (Meinck et al., 2018). The item will assess emotional abuse by asking parents/caregivers, "How many days in the past week did you shout, scream, or yell at your children?"
Change over time in Positive Parenting | Through study completion, an average of 16 weeks
  Positive parenting will be assessed two items from the Alabama Parenting Questionnaire (APQ) (Frick, 1991). The items included are "How many days in the past week did you and your child do something fun together?" and "How many days in the past week did you praise your child for doing well?" The parent/caregiver will be asked to give a frequency score, on a scale of 0 to 7 times.
Change over time in Parenting Stress | Through study completion, an average of 16 weeks
  Parenting stress will be assessed using one item adapted from the Parenting Stress Scale (PSS) (Berry & Jones, 1995). The item asks, "How many days in the past week did you feel very stressed as a parent/caregiver?" The items will be rated on a frequency scale of 0 to 7 times.
Change over time in Financial Stress | Through study completion, an average of 16 weeks
  Financial stress will be assessed using two items adapted from the Financial Self-Efficacy Scale (FSES) (Lown, 2011). The first items asks, "How many days in the past week have you felt very worried or anxious about money?" The parent/caregiver will be asked to give a frequency score, on a scale of 0 to 7 times. The second item asks, "How many days in the past month (30 days) did you run out of money to pay for food?" The parent/caregiver will be asked to indicate the number of days by typing a number between 0 and 30.
Change over time in Parental Self-efficacy | Through study completion, an average of 16 weeks
  Parental self-efficacy will be assessed using one item was adapted from the Parenting Sense of Competence Scale (Ohan et al., 2000). The item asks, "How confident do you feel about your ability as a parent/caregiver to have a positive relationship with your children? Parents/caregivers will respond based on an 8-point Likert scale of ranging from 0 (not confident) to 7 (extremely confident).
Change over time in Parental Communication about Sexual Abuse Prevention | Through study completion, an average of 16 weeks
  Parental Communication about Sexual Abuse Prevention will be assessed using two items adapted from the Parent Teen Sexual Risk Communication Scale III (PTSRC-III) (Hutchinson, 2007). One item asks, "In the past month, have you talked with your teen about keeping them safe from sexual violence in the community or online?" Parents/caregivers can respond yes or no. If they respond yes, they will be asked, "How many days have you had a talk like this?". The parent/caregiver will be asked to indicate the number of days by typing a number between 0 and 30.
Change over time in Child Behaviour Problems | Through study completion, an average of 16 weeks
  Child behaviour problems will be assessed using an adapted version of the Parent Daily Report (PDR) (Chamberlain & Reid, 1987). Parents/Caregivers are presented with a list of ten typical behaviours that can be challenging for parents that are relevant to their child's age groups. Parents/caregivers are asked to select the behaviour which describes the most challenging behaviours. Parents/caregivers are asked to indicate how challenging the chosen behaviour is on a scale of 0 to 7 (0 = not a problem, 7= terrible).
Change over time in Female IPV Victimisation | Through study completion, an average of 16 weeks and 1 and 3 months follow up
  Female IPV victimisation will be measured using items on physical violence (1 item), psychological abuse (1 item), sexual abuse (1 item), coercion (1 item), and economic abuse (1 item). Female IPV perpetration will be assessed using two items adapted from the VAWI (García-Moreno et al., 2005), which ask: "During any potential times that you were hit in the past month, did you ever fight back physically to defend yourself?" and "In the past month, have you ever hit or physically mistreated your partner when they were not hitting or physically mistreating you?". The female IPV assessment at baseline will also include one item that asks participants about any experiences of IPV victimisation they may have had in the past 12 months. Parents/caregivers are asked to give a frequency score on a scale of 0 to +8 times.
Change over time in Male IPV Perpetration | Through study completion, an average of 16 weeks and 1 and 3 months follow up
  Male IPV perpetration will be measured using items on physical violence (1 item), psychological abuse (1 item), sexual abuse (1 item), coercion (1 item), and economic abuse (1 item). Male IPV victimisation will be assessed using two items adapted from the VAWI: "In the past month, during any potential times that you may have used violence against your partner, did they ever fight back physically to defend themselves?" and "In the past month, have you ever been hit or physically mistreated by your partner when you were not hitting or physically mistreating them?". The male IPV assessment at baseline will also include one item that asks participants about any their experiences of IPV perpetration in the past 12 months. Parents/caregivers are asked to give a frequency score on a scale of 0 to +8 times.
Change over time in Attitudes towards gender roles and IPV | Through study completion, an average of 16 weeks and 1 and 3 months follow up
  Attitudes towards gender roles and IPV will be measured by self-report using six items included in the 'Attitudes toward gender roles' section of the WHO Multi-Country Study on Domestic Violence (García-Moreno et al., 2005). These items include statements such as "A woman should obey her husband's wishes even if she disagrees". . Parents/caregivers are asked to indicate whether they agree or disagree with the statements provided based on a Likert scale ranging from 1 (strongly agree) to 5 (strongly disagree).
Gender equitable behaviours | Through study completion, an average of 16 weeks and 1 and 3 months follow up
  Gender equitable behaviours will be measured using four items adapted from a questionnaire developed by researchers at the London School of Hygiene and Tropical Medicine which was used in an RCT of a violence prevention intervention in Tanzania (Kapiga et al., 2019). These items include questions on couple communication, joint decision-making, shared housework and caregiving, and partner conflict resolution, with questions such as: 'In the past week, how many times did you and your partner talk about your worries and feelings?" and "In the past week, how many times did you and your partner make a decision together?". Parents/caregivers are asked to report on whether in the past week the specific behaviour occurred on a scale of 0 (never) to 3 (many times).

OTHER OUTCOMES:
Demographics | Through study completion, an average of 16 weeks
  The parent/caregiver will be asked for their name, gender, and relationship status, country, state, as well as their relationship to the child, the child's name, gender, and age-group and age. They will also be asked if they are a parent/caregiver of a child living with disabilities.
Impact of COVID-19 | Through study completion, an average of 16 weeks
  Participants will be asked, how has COVID-19 affected their family? The participant will be asked to indicate one of the 6 options (someone in my family has had COVID-19 symptoms, someone in my family has died of COVID-19, my family has been experiencing financial stress due to COVID-19, family has been experiencing emotional stress due to COVID-19, my family has not been negatively affected by COVID-19, my family has not been affected by COVID-19). Participants will also be asked whether their children currently go to school/day-care?
Helpfulness of tips | Through study completion, an average of 16 weeks
  Participants will be asked, whether the advice was helpful? (Not helpful; A little helpful; helpful; very helpful; extremely helpful; prefer not to say). Participants will be asked whether the programme was helpful in improving their relationship with their child. Participants will also be asked which parenting tip they found the most useful.
Acceptability of the Programme | Through study completion, an average of 16 weeks
  Participants will be asked questions in regards to their experience with the programme. First participants will be asked to "tell us about the length of the ParentText programme (total number of days you received messages). ParentText was.. . 1)Too short, 2) Just right, 3) Too long. The second question asks participants "tell us about the number of messages that you received each day. They were... 1) Too few, 2) Just right, 3) Too many. Lastly, participants will also be asked an open-ended question, "Is there anything we can do to improve the ParentText chatbot for other families?".

CONTACTS AND LOCATIONS:
Overall Officials: Rumaya Binti Juhari, Dr, Principal Investigator — Universiti Putra Malaysia; Liane Peña Alampay, Dr, Principal Investigator — Ateneo de Manila University; Rosanne Jocson, Dr, Principal Investigator — Ateneo de Manila University; Hlengiwe Sacolo, Dr, Principal Investigator — University of Cape Town; Frances Gardner, Dr, Principal Investigator — University of Oxford; Joyce Wamoyi, Dr, Principal Investigator — Tanzania National Institute of Medical Research); Ytske Van Winden, Principal Investigator — UNICEF Jamaica; David Stern, Dr, Principal Investigator — IDEMS International
Locations (1):
- Family and Child Ecology at the Department of Human Development and Family Studies, Putrajaya, Putraja, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data will be shared on Open Science Framework after the completion of the study and once the results have been published.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Indefinitely
Access Criteria: Accessibility of the data will require approval from the study team. The study investigators, led by the PI, will jointly make decisions on whether to supply research data to potential new users. Research data will be deposited in and available in the UK Data Archive solely for non-profit use.

REFERENCES:
- [Background] Ariely, D., Bracha, A., & Meier, S. (2009). Doing Good or Doing Well? Image Motivation and Monetary Incentives in Behaving Prosocially. American Economic Review, 99(1), 544-555.
- [Background] Asbjornsen RA, Smedsrod ML, Solberg Nes L, Wentzel J, Varsi C, Hjelmesaeth J, van Gemert-Pijnen JE. Persuasive System Design Principles and Behavior Change Techniques to Stimulate Motivation and Adherence in Electronic Health Interventions to Support Weight Loss Maintenance: Scoping Review. J Med Internet Res. 2019 Jun 21;21(6):e14265. doi: 10.2196/14265. PMID 31228174
- [Background] Axford, N., Lehtonen, M., Kaoukji, D., Tobin, K., & Berry, V. (2012). Engaging parents in parenting programs: Lessons from research and practice. Children and Youth Services Review, 34(10), 2061-2071.
- [Background] Baker CN, Arnold DH, Meagher S. Enrollment and attendance in a parent training prevention program for conduct problems. Prev Sci. 2011 Jun;12(2):126-38. doi: 10.1007/s11121-010-0187-0. PMID 21052834
- [Background] Baumel A, Pawar A, Kane JM, Correll CU. Digital Parent Training for Children with Disruptive Behaviors: Systematic Review and Meta-Analysis of Randomized Trials. J Child Adolesc Psychopharmacol. 2016 Oct;26(8):740-749. doi: 10.1089/cap.2016.0048. Epub 2016 Jun 10. PMID 27286325
- [Background] Beatty L, Binnion C. A Systematic Review of Predictors of, and Reasons for, Adherence to Online Psychological Interventions. Int J Behav Med. 2016 Dec;23(6):776-794. doi: 10.1007/s12529-016-9556-9. PMID 26957109
- [Background] Berry, J. O., & Jones, W. H. (1995). The Parental Stress Scale - Initial Psychometric Evidence. Journal of Social and Personal Relationships, 12(3), 463-472.
- [Background] Braun, V., & Clarke, V. (2006). Using thematic analysis in psychology. Qualitative research in psychology, 3(2), 77-101.
- [Background] Burns, G. L., Lee, S., Servera, M., McBurnett, K., & Becker, S. P. (2015). Child and Adolescent Behavior Inventory - Version 1.
- [Background] Cacioppo, J. T., & Petty, R. E. (1989). Effects of message repetition on argument processing, recall, and persuasion. Basic and Applied Social Psychology, 10(1), 3-12.
- [Background] Chamberlain, P., & Reid, J. B. (1987). Parent observation and report of child symptoms. Behavioral Assessment.
- [Background] Cheong MWL, Allotey P, Reidpath DD. Unequal Access to Vaccines Will Exacerbate Other Inequalities. Asia Pac J Public Health. 2020 Sep-Oct;32(6-7):379-380. doi: 10.1177/1010539520944726. Epub 2020 Jul 25. No abstract available. PMID 32715721
- [Background] Collins LM, Murphy SA, Strecher V. The multiphase optimization strategy (MOST) and the sequential multiple assignment randomized trial (SMART): new methods for more potent eHealth interventions. Am J Prev Med. 2007 May;32(5 Suppl):S112-8. doi: 10.1016/j.amepre.2007.01.022. PMID 17466815
- [Background] Dadds MR, Sicouri G, Piotrowska PJ, Collins DAJ, Hawes DJ, Moul C, Lenroot RK, Frick PJ, Anderson V, Kimonis ER, Tully LA. Keeping Parents Involved: Predicting Attrition in a Self-Directed, Online Program for Childhood Conduct Problems. J Clin Child Adolesc Psychol. 2019 Nov-Dec;48(6):881-893. doi: 10.1080/15374416.2018.1485109. Epub 2018 Aug 1. PMID 30067388
- [Background] Daley K, Hungerbuehler I, Cavanagh K, Claro HG, Swinton PA, Kapps M. Preliminary Evaluation of the Engagement and Effectiveness of a Mental Health Chatbot. Front Digit Health. 2020 Nov 30;2:576361. doi: 10.3389/fdgth.2020.576361. eCollection 2020. PMID 34713049
- [Background] Dittman CK, Farruggia SP, Palmer ML, Sanders MR, Keown LJ. Predicting success in an online parenting intervention: the role of child, parent, and family factors. J Fam Psychol. 2014 Apr;28(2):236-243. doi: 10.1037/a0035991. Epub 2014 Mar 10. PMID 24611694
- [Background] Edney S, Ryan JC, Olds T, Monroe C, Fraysse F, Vandelanotte C, Plotnikoff R, Curtis R, Maher C. User Engagement and Attrition in an App-Based Physical Activity Intervention: Secondary Analysis of a Randomized Controlled Trial. J Med Internet Res. 2019 Nov 27;21(11):e14645. doi: 10.2196/14645. PMID 31774402
- [Background] Ellsberg, M., Heise, L., & Organization, W. H. (2005). Researching violence against women: a practical guide for researchers and activists.
- [Background] Falci SG, Marques LS. CONSORT: when and how to use it. Dental Press J Orthod. 2015 May-Jun;20(3):13-5. doi: 10.1590/2176-9451.20.3.013-015.ebo. No abstract available. PMID 26154451
- [Background] Florean IS, Dobrean A, Pasarelu CR, Georgescu RD, Milea I. The Efficacy of Internet-Based Parenting Programs for Children and Adolescents with Behavior Problems: A Meta-Analysis of Randomized Clinical Trials. Clin Child Fam Psychol Rev. 2020 Dec;23(4):510-528. doi: 10.1007/s10567-020-00326-0. Epub 2020 Sep 8. PMID 32897527
- [Background] Frick, P. J. (1991). The Alabama parenting questionnaire. Unpublished rating scale, University of Alabama.
- [Background] Garcia-Moreno C, Jansen HA, Ellsberg M, Heise L, Watts CH; WHO Multi-country Study on Women's Health and Domestic Violence against Women Study Team. Prevalence of intimate partner violence: findings from the WHO multi-country study on women's health and domestic violence. Lancet. 2006 Oct 7;368(9543):1260-9. doi: 10.1016/S0140-6736(06)69523-8. PMID 17027732
- [Background] Gonzalez C, Morawska A, Haslam DM. Enhancing Initial Parental Engagement in Interventions for Parents of Young Children: A Systematic Review of Experimental Studies. Clin Child Fam Psychol Rev. 2018 Sep;21(3):415-432. doi: 10.1007/s10567-018-0259-4. PMID 29611061
- [Background] Hackworth NJ, Matthews J, Westrupp EM, Nguyen C, Phan T, Scicluna A, Cann W, Bethelsen D, Bennetts SK, Nicholson JM. What Influences Parental Engagement in Early Intervention? Parent, Program and Community Predictors of Enrolment, Retention and Involvement. Prev Sci. 2018 Oct;19(7):880-893. doi: 10.1007/s11121-018-0897-2. PMID 29629506
- [Background] Hauser-Ulrich S, Kunzli H, Meier-Peterhans D, Kowatsch T. A Smartphone-Based Health Care Chatbot to Promote Self-Management of Chronic Pain (SELMA): Pilot Randomized Controlled Trial. JMIR Mhealth Uhealth. 2020 Apr 3;8(4):e15806. doi: 10.2196/15806. PMID 32242820
- [Background] Holt S, Buckley H, Whelan S. The impact of exposure to domestic violence on children and young people: a review of the literature. Child Abuse Negl. 2008 Aug;32(8):797-810. doi: 10.1016/j.chiabu.2008.02.004. Epub 2008 Aug 26. PMID 18752848
- [Background] Howick, J. (2011). Exposing the vanities-and a qualified defense-of mechanistic reasoning in health care decision making. Philosophy of Science, 78(5), 926-940.
- [Background] Hutchinson MK. The Parent-Teen Sexual Risk Communication Scale (PTSRC-III): instrument development and psychometrics. Nurs Res. 2007 Jan-Feb;56(1):1-8. doi: 10.1097/00006199-200701000-00001. PMID 17179868
- [Background] Jarvis, J. W., Gainforth, H. L., & Latimer-Cheung, A. E. (2014). Investigating the effect of message framing on parents' engagement with advertisements promoting child physical activity. International Review on Public and Nonprofit Marketing, 11(2), 115-127.
- [Background] Jenssen BP, Buttenheim AM, Fiks AG. Using Behavioral Economics to Encourage Parent Behavior Change: Opportunities to Improve Clinical Effectiveness. Acad Pediatr. 2019 Jan-Feb;19(1):4-10. doi: 10.1016/j.acap.2018.08.010. Epub 2018 Aug 30. PMID 30172918
- [Background] Kapiga S, Harvey S, Mshana G, Hansen CH, Mtolela GJ, Madaha F, Hashim R, Kapinga I, Mosha N, Abramsky T, Lees S, Watts C. A social empowerment intervention to prevent intimate partner violence against women in a microfinance scheme in Tanzania: findings from the MAISHA cluster randomised controlled trial. Lancet Glob Health. 2019 Oct;7(10):e1423-e1434. doi: 10.1016/S2214-109X(19)30316-X. PMID 31537372
- [Background] Katelin Wilton, M. S.C., Gabrielle Galanek & Katie Murphy. (2017). Parenting in Displacement, Adapting Vroom for Displacement.
- [Background] Klasnja P, Hekler EB, Shiffman S, Boruvka A, Almirall D, Tewari A, Murphy SA. Microrandomized trials: An experimental design for developing just-in-time adaptive interventions. Health Psychol. 2015 Dec;34S(0):1220-8. doi: 10.1037/hea0000305. PMID 26651463
- [Background] Kocielnik, R., & Hsieh, G. (2017). Send me a different message: utilizing cognitive space to create engaging message triggers. Proceedings of the 2017 ACM Conference on Computer Supported Cooperative Work and Social Computing.
- [Background] Knerr W, Gardner F, Cluver L. Improving positive parenting skills and reducing harsh and abusive parenting in low- and middle-income countries: a systematic review. Prev Sci. 2013 Aug;14(4):352-63. doi: 10.1007/s11121-012-0314-1. PMID 23315023
- [Background] Lehto, T., Oinas-Kukkonen, H., & Drozd, F. (2012). Factors affecting perceived persuasiveness of a behavior change support system.
- [Background] Leijten, P., Dishion, T. J., Thomaes, S., Raaijmakers, M. A., Orobio de Castro, B., & Matthys, W. (2015). Bringing parenting interventions back to the future: How randomized microtrials may benefit parenting intervention efficacy. Clinical psychology: science and practice, 22(1), 47-57.
- [Background] Levin C, Chisholm D. Cost-Effectiveness and Affordability of Interventions, Policies, and Platforms for the Prevention and Treatment of Mental, Neurological, and Substance Use Disorders. In: Patel V, Chisholm D, Dua T, Laxminarayan R, Medina-Mora ME, editors. Mental, Neurological, and Substance Use Disorders: Disease Control Priorities, Third Edition (Volume 4). Washington (DC): The International Bank for Reconstruction and Development / The World Bank; 2016 Mar 14. Chapter 12. Available from http://www.ncbi.nlm.nih.gov/books/NBK361929/ PMID 27227237
- [Background] Digolo, L. K. A., Rumble, L., Heise L., Berry V.L., Mitchell., S., & Alemann, C.(2019). EVIDENCE REVIEW: PARENTING AND CAREGIVER SUPPORT PROGRAMMES TO PREVENT AND RESPOND TO VIOLENCE IN THE HOME.
- [Background] Lown, J. M. (2011). Development and validation of a financial self-efficacy scale. Journal of Financial Counseling and Planning, 22(2), 54.
- [Background] McCoy A, Melendez-Torres GJ, Gardner F. Parenting interventions to prevent violence against children in low- and middle-income countries in East and Southeast Asia: A systematic review and multi-level meta-analysis. Child Abuse Negl. 2020 May;103:104444. doi: 10.1016/j.chiabu.2020.104444. Epub 2020 Mar 11. PMID 32171126
- [Background] Meinck F, Boyes ME, Cluver L, Ward CL, Schmidt P, DeStone S, Dunne MP. Adaptation and psychometric properties of the ISPCAN Child Abuse Screening Tool for use in trials (ICAST-Trial) among South African adolescents and their primary caregivers. Child Abuse Negl. 2018 Aug;82:45-58. doi: 10.1016/j.chiabu.2018.05.022. Epub 2018 May 31. PMID 29860107
- [Background] Metzler CW, Sanders MR, Rusby JC, Crowley RN. Using consumer preference information to increase the reach and impact of media-based parenting interventions in a public health approach to parenting support. Behav Ther. 2012 Jun;43(2):257-70. doi: 10.1016/j.beth.2011.05.004. Epub 2011 Jun 1. PMID 22440064
- [Background] Michie S, Yardley L, West R, Patrick K, Greaves F. Developing and Evaluating Digital Interventions to Promote Behavior Change in Health and Health Care: Recommendations Resulting From an International Workshop. J Med Internet Res. 2017 Jun 29;19(6):e232. doi: 10.2196/jmir.7126. PMID 28663162
- [Background] Network, B. C. (2020). The Alliance for Child Protection in Humanitarian Action, United Nations Children's Fund (UNICEF). Protection of children during the COVID-19 Pandemic, 2020-2005.
- [Background] Nøkleby, H., Flodgren, G. M., & Langøien, L. J. (2019). Digitale tiltak for foreldrestøtte: en systematisk oversikt over effekter og erfaringer.
- [Background] Ohan, J. L., Leung, D. W., & Johnston, C. (2000). The Parenting Sense of Competence scale: Evidence of a stable factor structure and validity. Canadian Journal of Behavioural Science/Revue canadienne des sciences du comportement, 32(4), 251.
- [Background] Orji R, Moffatt K. Persuasive technology for health and wellness: State-of-the-art and emerging trends. Health Informatics J. 2018 Mar;24(1):66-91. doi: 10.1177/1460458216650979. Epub 2016 May 31. PMID 27245673
- [Background] Patterson GR, Chamberlain P, Reid JB. A Comparative Evaluation of a Parent-Training Program -Republished Article. Behav Ther. 2016 Nov;47(6):804-811. doi: 10.1016/j.beth.2016.11.004. Epub 2016 Nov 10. PMID 27993334
- [Background] Pereda N, Diaz-Faes DA. Family violence against children in the wake of COVID-19 pandemic: a review of current perspectives and risk factors. Child Adolesc Psychiatry Ment Health. 2020 Oct 20;14:40. doi: 10.1186/s13034-020-00347-1. eCollection 2020. PMID 33088340
- [Background] Pereira J, Diaz O. Using Health Chatbots for Behavior Change: A Mapping Study. J Med Syst. 2019 Apr 4;43(5):135. doi: 10.1007/s10916-019-1237-1. PMID 30949846
- [Background] Perski O, Blandford A, West R, Michie S. Conceptualising engagement with digital behaviour change interventions: a systematic review using principles from critical interpretive synthesis. Transl Behav Med. 2017 Jun;7(2):254-267. doi: 10.1007/s13142-016-0453-1. PMID 27966189
- [Background] Runyan DK, Dunne MP, Zolotor AJ, Madrid B, Jain D, Gerbaka B, Menick DM, Andreva-Miller I, Kasim MS, Choo WY, Isaeva O, Macfarlane B, Ramirez C, Volkova E, Youssef RM. The development and piloting of the ISPCAN Child Abuse Screening Tool-Parent version (ICAST-P). Child Abuse Negl. 2009 Nov;33(11):826-32. doi: 10.1016/j.chiabu.2009.09.006. Epub 2009 Oct 24. PMID 19854511
- [Background] Ryan C, Bergin M, Wells JS. Theoretical Perspectives of Adherence to Web-Based Interventions: a Scoping Review. Int J Behav Med. 2018 Feb;25(1):17-29. doi: 10.1007/s12529-017-9678-8. PMID 28730402
- [Background] Ryan J, Edney S, Maher C. Engagement, compliance and retention with a gamified online social networking physical activity intervention. Transl Behav Med. 2017 Dec;7(4):702-708. doi: 10.1007/s13142-017-0499-8. PMID 28523603
- [Background] Sanders MR, Baker S, Turner KM. A randomized controlled trial evaluating the efficacy of Triple P Online with parents of children with early-onset conduct problems. Behav Res Ther. 2012 Nov;50(11):675-84. doi: 10.1016/j.brat.2012.07.004. Epub 2012 Aug 18. PMID 22982082
- [Background] Sanders MR, Dittman CK, Farruggia SP, Keown LJ. A comparison of online versus workbook delivery of a self-help positive parenting program. J Prim Prev. 2014 Jun;35(3):125-33. doi: 10.1007/s10935-014-0339-2. PMID 24500106
- [Background] Schuetzler, R. M., Grimes, G. M., & Scott Giboney, J. (2020). The impact of chatbot conversational skill on engagement and perceived humanness. Journal of Management Information Systems, 37(3), 875-900.
- [Background] Shi, W., Wang, X., Oh, Y. J., Zhang, J., Sahay, S., & Yu, Z. (2020). Effects of persuasive dialogues: testing bot identities and inquiry strategies. Proceedings of the 2020 CHI Conference on Human Factors in Computing Systems.
- [Background] Springer KW, Sheridan J, Kuo D, Carnes M. Long-term physical and mental health consequences of childhood physical abuse: results from a large population-based sample of men and women. Child Abuse Negl. 2007 May;31(5):517-30. doi: 10.1016/j.chiabu.2007.01.003. PMID 17532465
- [Background] Strecher VJ, Shiffman S, West R. Randomized controlled trial of a web-based computer-tailored smoking cessation program as a supplement to nicotine patch therapy. Addiction. 2005 May;100(5):682-8. doi: 10.1111/j.1360-0443.2005.01093.x. PMID 15847626
- [Background] Tippens KM, Chao MT, Connelly E, Locke A. Patient perspectives on care received at community acupuncture clinics: a qualitative thematic analysis. BMC Complement Altern Med. 2013 Oct 29;13:293. doi: 10.1186/1472-6882-13-293. PMID 24168022
- [Background] Tully LA, Piotrowska PJ, Collins DAJ, Mairet KS, Black N, Kimonis ER, Hawes DJ, Moul C, Lenroot RK, Frick PJ, Anderson V, Dadds MR. Optimising child outcomes from parenting interventions: fathers' experiences, preferences and barriers to participation. BMC Public Health. 2017 Jun 7;17(1):550. doi: 10.1186/s12889-017-4426-1. PMID 28592244
- [Background] Weisenmuller C, Hilton D. Barriers to access, implementation, and utilization of parenting interventions: Considerations for research and clinical applications. Am Psychol. 2021 Jan;76(1):104-115. doi: 10.1037/amp0000613. Epub 2020 Mar 5. PMID 32134281
- [Background] Werntz A, Bufka L, Adams BE, Teachman BA. Improving the reach of clinical practice guidelines: An experimental investigation of message framing on user engagement. Clin Psychol Sci. 2020 Sep 1;8(5):825-838. doi: 10.1177/2167702620920722. Epub 2020 Jul 2. PMID 33758685
- [Background] Widom, C. S. (2017). Long-term impact of childhood abuse and neglect on crime andviolence. Clinical psychology: science and practice, 24(2), 186-202.
- [Background] Yardley L, Spring BJ, Riper H, Morrison LG, Crane DH, Curtis K, Merchant GC, Naughton F, Blandford A. Understanding and Promoting Effective Engagement With Digital Behavior Change Interventions. Am J Prev Med. 2016 Nov;51(5):833-842. doi: 10.1016/j.amepre.2016.06.015. PMID 27745683
- [Background] Zeng Y, Guo Y, Li L, Hong YA, Li Y, Zhu M, Zeng C, Zhang H, Cai W, Liu C, Wu S, Chi P, Monroe-Wise A, Hao Y, Ho RTH. Relationship Between Patient Engagement and Depressive Symptoms Among People Living With HIV in a Mobile Health Intervention: Secondary Analysis of a Randomized Controlled Trial. JMIR Mhealth Uhealth. 2020 Oct 29;8(10):e20847. doi: 10.2196/20847. PMID 33118956
- [Background] Zhu M, Cai W, Li L, Guo Y, Monroe-Wise A, Li Y, Zeng C, Qiao J, Xu Z, Zhang H, Zeng Y, Liu C. Mediators of Intervention Effects on Depressive Symptoms Among People Living With HIV: Secondary Analysis of a Mobile Health Randomized Controlled Trial Using Latent Growth Curve Modeling. JMIR Mhealth Uhealth. 2019 Nov 15;7(11):e15489. doi: 10.2196/15489. PMID 31730042